CLINICAL TRIAL: NCT00447746
Title: A Comparison Between D1 and D2 Lymphadenectomy in Gastric Cancer : A Prospective Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMH 262
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Gastric Cancer
Keywords: Comparison between D1 and D2 lymphadenectomy for gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: D1 or D2 lymphadenectomy for gastric cancer patients

SUMMARY:
Gastric cancer remains the second most common cancer worldwide.Although the prognosis is poor for majority of patients , long term survival is achievable in patients in whom surgical resection is possible.

However the results of surgery are generally disapointing in most large series.The exception to this appears to be Japan and far east where a standardized approach to surgery is undertaken with low morbidity and mortality.The extent of surgery and particularly the development of systematic lymphadenectomy(D2)has been credited in Japan for the improved outcome in patients with gastric cancer.

Hence for comparing the difference between D1 and D2 lymphadenectomy for gastric cancer in terms of overall survival,disease free survival and loco regional recurrence and also post operative morbidity and mortality following both these procedures,this study has been undertaken.

In D1 lymphadenectomy, only those lymph nodes which are adjacent to the part of stomach being resected will be removed.In D2 lymphadenectomy other lymph nodes draining the stomach will also be removed according to internationally accepted guidelines and also include resection of greater omentum along with anterior layer of transverse mesocolon and lesser omentum upto its attachment to hepatoduodenal ligament.

Currently both these procedures are widely practised worldwide and there is no definite evidence showing the superiority of one procedure over the other.Neither is any of these procedures experimental.

We are doing this trial to see whether one of these procedures is superior to the other.

ELIGIBILITY:
Inclusion Criteria:Patients with biopsy/frozen section proven adenocarcinoma of stomach.

* Preoperative clinical examination and imaging indicating operable disease.
* Intraoperative exploration indicating operability i.e. no peritoneal deposits,no evidence of para aortic lymphadenopathy,no direct involvement of contiguous organs
* Surgical plan for distal/proximal/total gastrectomy

Exclusion Criteria:Patients with low performance score

* Staging investigations or intraoperative exploration indicating inoperable disease
* Patients medically unfit for major surgery
* Patients who have been given preoperative chemotherapy/chemoradiation.
* Patients with gastroesophageal junction tumours
* Patients unreliable for follow up
* Patients above the age of 70 years
* Past history of malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2007-03; Study Completion 2014-03

PRIMARY OUTCOMES:
5 year overall survival

SECONDARY OUTCOMES:
: 5 year disease free survival
: 5 year local recurrence
: Postoperative morbidity and mortality rates

CONTACTS AND LOCATIONS:
Overall Officials: Dr Parul J Shukla, M.S.,FRCS, Principal Investigator — Tata Memorial Centre,Mumbai
Locations (1):
- Tata Memorial Hospital,Tata Memorial Centre, Mumbai, Maharashtra, India